CLINICAL TRIAL: NCT03201887
Title: Detecting Malingering Detection Using Eye Movements and Response Time
Brief Title: Detecting Malingering Detection Using Eye Movements and Response Time (MDER)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Loewenstein Hospital (Other)
Collaborators: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Tasmc16ys0ctil
Record Dates: First submitted 2017-01-17; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-01

CONDITIONS: Traumatic Brain Damage; Chronic Pain
MeSH Terms: conditions — Brain Injuries, Traumatic; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sub-optimal Traumatic Brain Injury (Experimental): Sub-optimal effort
  Interventions: Behavioral: Sub-optimal effort; Behavioral: optimal effort
- Sub-optimal effort Chronic pain (Experimental): Sub-optimal effort
  Interventions: Behavioral: Sub-optimal effort; Behavioral: optimal effort
- Traumatic Brain Injury (No Intervention): optimal effort
- Chronic pain (No Intervention): optimal effort

INTERVENTIONS:
Behavioral: Sub-optimal effort — Participants will be asked to play a patient who wishes to present himself as having cognitive deficits or exaggerate existing cognitive deficits
  Other Names: Simulation condition
  Arms: Sub-optimal Traumatic Brain Injury; Sub-optimal effort Chronic pain
Behavioral: optimal effort — Participants will be asked to perform tasks to the best of their abilities.
  Other Names: control condition
  Arms: Sub-optimal Traumatic Brain Injury; Sub-optimal effort Chronic pain

SUMMARY:
Performance Validity Tests (PVTs) are widely used for the detection of sub-optimal effort and malingering in neuropsychological assessments. Threats to their validity however likely to intensify with time (e.g., information available on the web or from legal representatives) and may lead to a decline in their ability to differentiate between malingerers and non-malingerers. Eye movements and response time (RT) are less obvious outcome measures and under less conscious control than more conventional PVT indices (e.g., accuracy). They are therefore promising measures that can aid in detecting malingering when used in conjunction with more conventional PVT indices. The Word Memory Test (WMT) is a widely used PVT in neuropsychological evaluations. As part of the proposed study, TBI patients, chronic pain patients and healthy adults (60 in each group) will be randomly divided to one of two conditions; optimal effort or sub-optimal effort (participants will be asked to play a TBI patient who wishes to present himself as having cognitive deficits or exaggerate existing cognitive deficits). The proposed study will improve the WMT's efficacy in detection of sub-optimal effort in neuropsychological evaluations and therefore protect its validity from future threats. In addition, the proposed study will provide us with better understanding of the effect of TBI on eye movements and RTs in general.

DETAILED DESCRIPTION:
Same as in the brief summary

ELIGIBILITY:
Inclusion criteria for all participants:

* Adult (18-65) female and males.
* Signed informed consent form.

Inclusion criteria for TBI group:

* TBI of at least mild severity, as operationalized by Post traumatic amnesia (PTA) < 24 hours
* Glasgow coma scale (GCS) of 13-15
* Loss of consciousness (LOC) of 30 minutes or less.

Inclusion criteria for chronic pain patients:

• Pain without apparent biological value that has persisted beyond three months. This will be based on the participant self-report, electronic medical records and consultation with treating physician.

Exclusion Criteria:

- Exclusion criteria for all participants:

* Any current eye impairment (e.g., limited visual field, nystagmus, astigmatism [cylinder], strabismus or any other impairment specified by the participant), past strabismus, and refractive surgery.
* Significant past neurological disorder/s and/or neurosurgery (special emphasis will be put on any language impairment such as aphasia).
* Significant developmental disorders (e.g., learning disabilities such as dyslexia). (d)
* Significant past or present psychiatric disorders (as evident, for example, in psychiatric inpatient hospitalization and past suicide attempts).
* Exclusion according to the last three articles (a-c) will be decided by a joint consultation of the research team.
* Exclusion criteria for TBI patients and healthy adults:
* Any condition of chronic pain (see criteria in the inclusion for the chronic pain group).
* Exclusion criteria for chronic pain patients and health adults:
* Significant current neurological disorder/s (special emphasis will be put on any language impairment such as aphasia) as decided by a joint consultation of the research team.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Eye Movements | 1 month
  Eye tracking used to evaluate eye behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Moti Ratmansky, MD, Principal Investigator — Loewenstein Hospital

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD